CLINICAL TRIAL: NCT03397680
Title: Effectiveness of Once-daily Dose Regimen of 7-day and 14-day High Dose Rabeprazole-levofloxacin Based Quadruple Therapy for H. Pylori Eradication in Thai Patients With Non-ulcer Dyspepsia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Jeerayuth Auttajaroon, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-IM-2-200/59
Record Dates: First submitted 2017-09-09; First posted 2018-01-12 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori infection; Non-ulcer Dyspepsia; Rabeprazole-Levofloxacin

STUDY DESIGN:
Intervention Model Description: Participants with positive rapid urease test or pathologic findings were divided into 2 groups and enrolled into randomization with 1:1 block of four methods. Each participant in group1 received 7-day once daily dose regimen of 1-tablet 750-mg Levofloxacin after meal, 2-tablet 500-mg Clarithromycin MR after meal, 3-tablet 20-mg Rabeprazole before meal and 1-tablet 1,048-mg Gastro bismol after meal.
  Meanwhile, each participant in group2 received 14-day once daily dose regimen of 1-tablet 750-mg Levofloxacin after meal, 2-tablet 500-mg Clarithromycin MR after meal, 3-tablet 20-mg Rabeprazole before meal and 1-tablet 1,048-mg Gastro bismol after meal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rabeprazole-levofloxacin based quadruple therapy for 7 days (Active Comparator): Participant will received 7-day once daily dose regimen of 1-tablet 750-mg Levofloxacin after meal, 2-tablet 500-mg Clarithromycin MR after meal, 3-tablet 20-mg Rabeprazole before meal and 1-tablet 1,048-mg Gastro bismol after meal.
  Interventions: Diagnostic Test: 13C Urea Breath Test
- Rabeprazole-levofloxacin based quadruple therapy for14 days (Active Comparator): Pparticipant will received 14-day once daily dose regimen of 1-tablet 750-mg Levofloxacin after meal, 2-tablet 500-mg Clarithromycin MR after meal, 3-tablet 20-mg Rabeprazole before meal and 1-tablet 1,048-mg Gastro bismol after meal
  Interventions: Diagnostic Test: 13C Urea Breath Test

INTERVENTIONS:
Diagnostic Test: 13C Urea Breath Test — After the H.pylori eradication treatment course completed, participants then was tested with 13C Urea Breath Test to confirm treatment effectiveness at least after ceasing PPI and antibiotics for 4 weeks.

SUMMARY:
H.pylori is an organism which causes gastric inflammation, peptic ulcer disease (PUD), mucosa associated lymphoid tissue (MALT) lymphoma and gastric cancer.

Practical guideline for treatment of patients with dyspepsia and H.pylori eradication recommended the 14-day triple therapy regimen which had curable about 70% by using proton pump inhibitor (PPI) combined with antibiotics including amoxicillin, clarithromycin and metronidazole.

Up to date, there has been no evidence about the cure rate for H.pylori eradication with once-daily dose regimen of high dose rabeprazole and levofloxacin based therapy. This research is to study the 7-day and 14-day cure rate of H.pylori eradication treatment with once-daily regimen of high dose rabeprazole-levofloxacin based quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Thai patients with the age between 18 and 70 years
* Detecting for H.pylori infection with positive urease test and/or pathological findings of H.pylori and/or positive

Exclusion criteria:

1. Any cases with upper gastrointestinal bleeding
2. Being treated with medications affecting the research outcome, for example, by using antibiotics including amoxicillin, clarithromycin, metronidazole or fluoroquinolone within 1 month before the enrollment.
3. Contraindicated for gastric biopsy such as coagulopathy.
4. Any history of drug allergy for levofloxacin, clarithromycin or rabeprazole.
5. Receiving proton pump inhibitor within 4 weeks or receiving any antibiotics or bismuth within 2 weeks.
6. Being pregnant or raising children with lactation.
7. Having history of H.pylori eradication treatment.
8. Having severe underlying disease including end-stage renal disease requiring hemodialysis or peritoneal dialysis (GFR < 15), cirrhosis with Child-Pugh classification grade C, immunocompromised host with AIDS, malignancy and/or bed ridden cerebrovascular disease.
9. Any cases who receiving anticoagulant.
10. Having previous gastric surgery.
11. Unwilling to participate into research.
12. Having history of taking previous medications which interacted with the research treatment.
13. Having underlying heart disease including congenital long QT syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-15 (Estimated)

PRIMARY OUTCOMES:
To measure eradication rate of participants with once-daily dose regimen of 14-day rabeprazole-levofloxacin based quadruple therapy for H. pylori eradication by Urea Breath Test in Thai patients with non-ulcer dyspepsia | 6 weeks
  Participants with positive rapid urease test or pathologic findings evidenced for H.pylori received 14-day once daily dose regimen. After the H.pylori eradication treatment course completed, participants then was tested with 13C Urea Breath Test to confirm the effectiveness of the treatment at 4 weeks. Eradication rate was defined as proportion of post-treatment cases with negative urea breath test compared to pre-treatment cases with positive rapid urease test or pathologic findings evidenced for H.pylori.
To measure eradication rate of participants with once-daily dose regimen of 7-day rabeprazole-levofloxacin based quadruple therapy for H. pylori eradication by Urea Breath Test in Thai patients with non-ulcer dyspepsia | 5 weeks
  Participants with positive rapid urease test or pathologic findings evidenced for H.pylori received 7-day once daily dose regimen. After the H.pylori eradication treatment course completed, participants then was tested with 13C Urea Breath Test to confirm the effectiveness of the treatment at 4 weeks. Eradication rate was defined as proportion of post-treatment cases with negative urea breath test compared to pre-treatment cases with positive rapid urease test or pathologic findings evidenced for H.pylori.

SECONDARY OUTCOMES:
To measure the adverse effect reaction of once-daily regimen of high dose rabeprazole-levofloxacin based quadruple therapy | up to 1 month
  To measure the adverse effect reaction up to 1 month after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Ratha-korn Vilaichone, Principal Investigator — Gastroenterology Unit, Department of Medicine, Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Khlong Luang, Patumthanee, Thailand

IPD SHARING:
Plan to Share IPD: Undecided